CLINICAL TRIAL: NCT00273832
Title: Randomized Controlled Trial of Multi-Slice Coronary Computed Tomography for Evaluation of Acute Chest Pain
Brief Title: Study of Coronary Artery Computed Tomography to Diagnose Emergency Chest Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Corewell Health East (Other)
Collaborators: The Minestrelli Advanced Cardiac Research Imaging Center, Royal Oak, Michigan (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: HIC - 2005 - 010
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Last update posted 2006-01-09 (Estimated); Status verified 2005-12

CONDITIONS: Chest Pain; Angina Pectoris; Myocardial Infarction
Keywords: Chest pain; Angina pectoris; Emergency medicine; Spiral computed tomography; Length of stay; Cost analysis
MeSH Terms: conditions — Chest Pain; Angina Pectoris; Myocardial Infarction

INTERVENTIONS:
Procedure: coronary artery computed tomography angiogram
Procedure: single photon emission computed tomography

SUMMARY:
The purpose of this study is to determine whether coronary artery computed tomography scanning is a more rapid, less expensive and safe alternative to standard diagnostic evaluation of patients with acute chest pain in the emergency room.

DETAILED DESCRIPTION:
Over 6 million patients per year visit hospital emergency departments for evaluation of chest pain, with diagnostic costs estimated to be in excess of $10 billion. Standard diagnostic evaluation often includes 8-12 hours of serial laboratory tests followed by stress imaging studies requiring an additional 4-8 hours.

Multi-slice coronary artery computed tomography scanning (MSCT) has been shown to be a highly accurate diagnostic method in comparison to invasive angiography. Because of its speed and high negative predictive value, MSCT could rapidly screen patients for the presence of coronary disease, which may expedite their care.

This study compares the length of stay and cost of care in emergency chest pain patients randomly assigned to initial evaluation by MSCT compared to patients randomly assigned to a standard diagnostic evaluation including single photon emission computed tomography scanning. The study follows these patients to detect major adverse cardiac events including unstable angina, acute myocardial infarction or death over a 90-day period.

ELIGIBILITY:
Inclusion Criteria:

* Chest pain or angina equivalent symptoms.
* Age ≥ 25 years.
* Low risk of infarction and/or complications by Goldman/Reilly criteria.

Exclusion Criteria:

* Known coronary artery disease.
* Electrocardiogram diagnostic of acute cardiac ischemia and/or infarction.
* Elevated serum biomarkers including creatine kinase (CK) MB, myoglobin, and/or cardiac troponin I on initial testing.
* Contraindication to iodinated contrast and/or beta blocking drugs.
* Atrial fibrillation or markedly irregular rhythm.
* Pregnancy.
* Renal insufficiency, creatinine > 1.5 mg/dL.
* Iodinated contrast within prior 48 hours.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2005-03; Study Completion 2005-11

PRIMARY OUTCOMES:
Length of stay
Cost of care

SECONDARY OUTCOMES:
Unstable angina within 90-days
Acute myocardial infarction within 90-days
Cardiac death within 90-days

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert L Raff, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

REFERENCES:
- [Background] Farkouh ME, Smars PA, Reeder GS, Zinsmeister AR, Evans RW, Meloy TD, Kopecky SL, Allen M, Allison TG, Gibbons RJ, Gabriel SE. A clinical trial of a chest-pain observation unit for patients with unstable angina. Chest Pain Evaluation in the Emergency Room (CHEER) Investigators. N Engl J Med. 1998 Dec 24;339(26):1882-8. doi: 10.1056/NEJM199812243392603. PMID 9862943
- [Background] Braunwald E, Antman EM, Beasley JW, Califf RM, Cheitlin MD, Hochman JS, Jones RH, Kereiakes D, Kupersmith J, Levin TN, Pepine CJ, Schaeffer JW, Smith EE 3rd, Steward DE, Theroux P, Gibbons RJ, Alpert JS, Faxon DP, Fuster V, Gregoratos G, Hiratzka LF, Jacobs AK, Smith SC Jr; American College of Cardiology; American Heart Association. Committee on the Management of Patients With Unstable Angina. ACC/AHA 2002 guideline update for the management of patients with unstable angina and non-ST-segment elevation myocardial infarction--summary article: a report of the American College of Cardiology/American Heart Association task force on practice guidelines (Committee on the Management of Patients With Unstable Angina). J Am Coll Cardiol. 2002 Oct 2;40(7):1366-74. doi: 10.1016/s0735-1097(02)02336-7. No abstract available. PMID 12383588
- [Background] Raff GL, Gallagher MJ, O'Neill WW, Goldstein JA. Diagnostic accuracy of noninvasive coronary angiography using 64-slice spiral computed tomography. J Am Coll Cardiol. 2005 Aug 2;46(3):552-7. doi: 10.1016/j.jacc.2005.05.056. PMID 16053973
- [Background] Zalenski RJ, Rydman RJ, Ting S, Kampe L, Selker HP. A national survey of emergency department chest pain centers in the United States. Am J Cardiol. 1998 Jun 1;81(11):1305-9. doi: 10.1016/s0002-9149(98)00159-3. PMID 9631967
- [Derived] Goldstein JA, Gallagher MJ, O'Neill WW, Ross MA, O'Neil BJ, Raff GL. A randomized controlled trial of multi-slice coronary computed tomography for evaluation of acute chest pain. J Am Coll Cardiol. 2007 Feb 27;49(8):863-71. doi: 10.1016/j.jacc.2006.08.064. Epub 2007 Feb 12. PMID 17320744